CLINICAL TRIAL: NCT04229329
Title: The Effect of Intensive Training on Recovery of Fingers Dexterity Following Stroke: Behavioral, Physiological and Anatomical Predictors
Brief Title: Effects of Intensive Training on Reocvery of Fingers Dexterity Following Stroke
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Nachum Soroker, MD, Head of Research, Department of Neurological Rehabilitation, Loewenstein Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LOE-19-19
Record Dates: First submitted 2019-12-31; First posted 2020-01-18 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The patient hand will be restrained to a robotic arm AMADEO(TM) which enables the measurement and manipulation of forces at each finger individually. After appropriate calibration, the force measurements obtained from the robot will be used to move a cursor on the screen. The patient will be rewarded visually and auditory when a higher degree of finger individuation will be measured. Specifically, when the applied force of the instructed fingers hit the predefined force target and at the same, the force in the non-instructed fingers stay as low as possible
  Interventions: Combination Product: Intensive Finger Individuation Therapy
- Control (Sham Comparator): The patient hand will be restrained to a robotic arm AMADEO(TM) which enables the measurement and manipulation of forces at each finger individually. After appropriate calibration, the force measurements obtained from the robot will be used to move a cursor on the screen. The patient will be rewarded in a way that is unrelated to the degree of individuation. In other words, a successful trial considered when the applied force of the instructed fingers hits the predefined force target regardless of the force exerted in the non-instructed fingers.
  Interventions: Combination Product: Intensive non-directed finger movement therapy

INTERVENTIONS:
Combination Product: Intensive Finger Individuation Therapy — Interactive robot-mediated treatment aimed at increased individuation done repeatedly for at least1 hour per day for 2 weeks (5 training days a week).
  Arms: Intervention
Combination Product: Intensive non-directed finger movement therapy — Interactive robot-mediated treatment not aimed specifically at increased individuation done repeatedly for at least 1 hour per day for 2 weeks (5 training days per week)
  Arms: Control

SUMMARY:
The investigators aim to test whether intensive training of finger individuation during the sensitive window of the subacute phases can lead to a clinically-meaningful recovery of dexterous movement in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* First symptomatic ischemic or hemorrhagic stroke
* Clinically evident upper-limb motor deficit
* Understand the study aim, is able to cooperate with the task for the specified time
* Clinically stable

Exclusion Criteria:

* Other neurological or psychiatric illness which affects upper-limb motor function
* An orthopedic or rheumatologic disease that affects the ability to undergo a robotic hand therapy.
* Sensory problems that prevent the patient from reporting pain during the robotic hand therapy
* Skin breakdown or wounds located in places where the hand contacts the robot.
* Patients with C/I to TMS (history of seizures, the existence of cardiac pacer, VP shunt, spinal stimulator or any other hardware that may malfunction at the presence of strong magnetic fields) will no undergo TMS but may participate in the study
* Participation in another interventional study for upper limb rehabilitation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment Score for Upper Extremity at the immediate post-intervention time | Change from Baseline Score at 1-3 days post-intervention
  A Likert-scale that quantifies movement quality, sensation, range of motion and pain in the upper limb following stroke. Range: 0 - 66. Higher values correlate with better motor control.
Change in Fugl-Meyer Assessment Score for Upper Extermity at 1-month post-intervention | Change from Baseline Score at 1 month post-intervention
  A Likert-scale that quantifies movement quality, sensation, range of motion and pain in the upper limb following stroke. Range: 0 - 66. Higher values correlate with better motor control.
Change in Fugl-Meyer Assessment Score for Upper Extermity at 3-month post-intervention | Change from Baseline Score at 3 month post-intervention
  A Likert-scale that quantifies movement quality, sensation, range of motion and pain in the upper limb following stroke. Range: 0 - 66. Higher values correlate with better motor control.
Change in Individuation Index at the immediate post-intervention time | Change from Baseline Score at 1-3 days post-intervention
  The relationship between forces (in Newton) in the active vs. passive fingers during a set of isolated finger movements. Higher numbers correlate with better finger-joint individuation, thus better dexterity.
Change in Individuation Index at 1-month post-intervention | Change from Baseline Score at 1-month post-intervention
  The relationship between forces (in Newton) in the active vs. passive fingers during a set of isolated finger movements. Higher numbers correlate with better finger-joint individuation, thus better dexterity.
Change in Individuation Index at 3-month post-intervention | Change from Baseline Score at 3-month post-intervention
  The relationship between forces (in Newton) in the active vs. passive fingers during a set of isolated finger movements. Higher numbers correlate with better finger-joint individuation, thus better dexterity.

SECONDARY OUTCOMES:
Arm Research Action Test (ARAT) Score at the immediate post-intervention time | Change from Baseline Score at 1-3 days post-intervention
  Time and quality of performance of 19 items mimicking activity of daily living, are measured. Tange: 0 - 57. Higher values correlate with better motor control.
Arm Research Action Test (ARAT) Score at at 1-month post-intervention | Change from Baseline Score at 1-month post-intervention
  Time and quality of performance of 19 items mimicking activity of daily living, are measured. Range: 0 - 57. Higher values correlate with better motor control.
Arm Research Action Test (ARAT) Score at at 3-month post-intervention | Change from Baseline Score at 3-month post-intervention
  Time and quality of performance of 19 items mimicking activity of daily living, are measured. Range: 0 - 57. Higher values correlate with better motor control.
Change in M1 MEP (motor evoked potentials) amplitude at immediate post-intervention time | Change from Baseline Score at 1-3 days post-intervention
  Stimulation of the ipsilesional M1 will be done (using either figure-of-eight, H- or dual-H rotational field coil) connected to TMS to elicit motor-evoked potential (MEP) of the first dorsal interosseous (FDI) muscle of the right hand, recorded with an EMG electrode. The peak-to-peak time will be computed off-line using MATLAB software. Higher MEP amplitudes correlate with higher cortico-spinal integrity.
Change in M1 MEP (motor evoked potentials) amplitude at 1-month post-intervention | Change from Baseline Score at 1-month post-intervention
  Stimulation of the ipsilesional M1 will be done (using either figure-of-eight, H- or dual-H rotational field coil) connected to TMS to elicit motor-evoked potential (MEP) of the first dorsal interosseous (FDI) muscle of the right hand, recorded with an EMG electrode. The peak-to-peak time will be computed off-line using MATLAB software. Higher MEP amplitudes correlate with higher cortico-spinal integrity.
Change in MEP (motor evoked potentials) amplitude at 3-months post-intervention | Change from Baseline Score at 3-months post-intervention
  Stimulation of the ipsilesional M1 will be done (using either figure-of-eight, H- or dual-H rotational field coil) connected to TMS to elicit motor-evoked potential (MEP) of the first dorsal interosseous (FDI) muscle of the right hand, recorded with an EMG electrode. The peak-to-peak time will be computed off-line using MATLAB software. Higher MEP amplitudes correlate with higher cortico-spinal integrity.
Change in extent of SICI (short-interval cortical inhibition) at the immediate post-intervention time | Change from Baseline Score at 1-3 days post-intervention
  Single test pulses, conditioning pulses (five of each) and paired pulses (five pairs) at an inter-stimuli-interval (ISI) of 2 ms will be delivered to the motor cortex of both hemispheres. The intensity of the conditioning stimulus will be set at 80% of the subject's resting motor threshold (MT). The intensity of the test pulse will be 110% of the resting MT. The SICI will be measured as the reduction in conditioned MEPs relative to baseline MEPs. Higher SICI correlates with increased inhibitory activity of the motor cortex.
Change in extent of SICI (short-interval cortical inhibition) at 1-month post-intervention | Change from Baseline Score at 1-month post-intervention
  Single test pulses, conditioning pulses (five of each) and paired pulses (five pairs) at an inter-stimuli-interval (ISI) of 2 ms will be delivered to the motor cortex of both hemispheres. The intensity of the conditioning stimulus will be set at 80% of the subject's resting motor threshold (MT). The intensity of the test pulse will be 110% of the resting MT. The SICI will be measured as the reduction in conditioned MEPs relative to baseline MEPs. Higher SICI correlates with increased inhibitory activity of the motor cortex.
Change in extent of SICI (short-interval cortical inhibition) at 3-months post-intervention | Change from Baseline Score at 3-months post-intervention
  Single test pulses, conditioning pulses (five of each) and paired pulses (five pairs) at an inter-stimuli-interval (ISI) of 2 ms will be delivered to the motor cortex of both hemispheres. The intensity of the conditioning stimulus will be set at 80% of the subject's resting motor threshold (MT). The intensity of the test pulse will be 110% of the resting MT. The SICI will be measured as the reduction in conditioned MEPs relative to baseline MEPs. Higher SICI correlates with increased inhibitory activity of the motor cortex.

CONTACTS AND LOCATIONS:
Locations (1):
- Loewenstein Rehabilitation Center, Raanana, Israel